CLINICAL TRIAL: NCT04558489
Title: Bridging the Gap: Utility of a Single Session Intervention to Change Attitudes Toward Treatment, and Improve Acceptance of Further Psychotherapy for Depressed and/or Anxious Youth and Their Caretakers
Brief Title: Bridging the Gap to Improve Mental Health Treatment Utilization
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study has withdrawn due to recruitment issues at our pediatric primary care setting. Due to the COVID-19 pandemic and other unforeseen medical absences, the study was unable to recruit participants.
Sponsor: University of Pittsburgh (Other)
Collaborators: Kaiser Foundation Research Institute (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Tina R Goldstein, Associate Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY19110071; P50MH115838-02 (NIH)
Record Dates: First submitted 2020-09-09; First posted 2020-09-22 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Depression; Anxiety; Adolescent Behavior; Suicidal Ideation
Keywords: depression; pediatric primary care; adolescent behavior; mood disorder; technology; provider; intervention
MeSH Terms: conditions — Depression; Anxiety Disorders; Adolescent Behavior; Suicidal Ideation; Mood Disorders

STUDY DESIGN:
Intervention Model Description: This study will use an open trial design, where all participants will receive the Growth Mindset Intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IPR + GMI (Experimental): Participants receiving IPR + GMI will complete a 30-minute on-line intervention via qualtrics that covers the following topics: (1) Educate youth and caregiver that thoughts and emotions are not fixed but are malleable and subject to change; (2) provide youth and families with a brief intervention that instills hopefulness through an action plan for managing internalizing symptoms; (3) assist with developing system of support to access during times of distress; and (4) educate the caregiver on the importance of these interventions.
  Interventions: Behavioral: IPR + GMI

INTERVENTIONS:
Behavioral: IPR + GMI — The IPR + GMI intervention aims to impact reported hopelessness, attitudes to treatment, and view of self as changeable as well as targets treatment attendance and utilization.

SUMMARY:
Bridging the Gap aims to improve access to effective mental health treatment in a primary care setting through utilization of single session growth mindset interventions for parents and for youths. This project will also utilize focus groups and qualitative interviews to gain feedback on a single session online intervention in a rural pediatric primary care practice.

DETAILED DESCRIPTION:
Bridging the Gap purposes to collect feedback on a single session growth mindset intervention (GMI) for parents and for youths designed to instill beliefs that personal traits (including mental health problems) are malleable. Feedback will also be collected to identify ways to improve implementing single session interventions (SSIs) in a primary care setting as well as identifying the impact on work-flow of this GMI. Patients presenting with depression and/or anxiety will all receive the GMI and will have the option of participating in focus groups/interviews pre and post-intervention to provide feedback on the intervention. Providers at this rural pediatric primary care practice will also have the chance to participate in focus groups/interviews pre and post-intervention implementation.

Assignment of Interventions: As an open trial, all participants will be assigned to the intervention arm and will receive the GMI.

This study is an open trial pilot project to collect feedback on a single session growth mindset intervention (GMI) (n=25 youth/caretaker dyads). Feedback from pre and post-intervention focus groups/interviews will be collected for 8 parents, 8 youth, and 8 treatment providers.

The aims of the study are to:

1. Collect feedback from providers, parents, and participants pre and post- GMI to identify ways to improve implementing single session interventions (SSIs) in a primary care setting.
2. Identify the impact on work-flow of using an online single session called Growth Mindset Intervention in a primary care setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with depression and/or anxiety, as identified by the patient, parent, or provider
* 10-18 years old
* CBT is recommended by provider. Receipt of mental health services upon enrollment will be monitored but will not preclude participation
* Participants must reside with a legal guardian
* English speaking

Exclusion Criteria:

* Participants will be excluded if they have conditions that might impair their ability to effectively engage in Bridging the Gap, i.e
* Those in a current manic episode
* Those in a current psychotic episode
* Those diagnosed with Autism Spectrum Disorder
* Those who have issues with substance abuse
* Participants with current involvement with child welfare.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-30 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in child and parental attitudes towards therapy at 4 weeks | Baseline vs. 4 week follow-up
  Child and parental attitudes towards therapy will be assessed via Attitudes Towards Therapy Scale, as the primary outcome of Bridging the Gap. Scores on this one question assessment range from 0= view of therapy as not at all helpful to 10= view of therapy as very helpful.
Change from baseline in view of emotions as changeable at 4 weeks | Baseline vs. 4 week follow-up
  Child and parental views of personality as changeable will be assessed via Implicit Theory of Emotions Scale, as the primary outcome of Bridging the Gap. The Implicit Theory of Emotion contains 4 questions, with two incremental items and two entity items. Each item is rated using a 7-point Likert scale with 1= strongly disagree and 7= strongly agree. The two entity items are reverse-scored. Scores range from 4-28 and higher scores indicate a view of emotions as changeable.
Change from baseline in view of personality as changeable at 4 weeks | Baseline vs. 4 week follow-up
  Child and parental views of personality as changeable will be assessed via Implicit Theory of Personality Questionnaire, as the primary outcome of Bridging the Gap. The Implicit Theory of Personality Questionnaire contains 3 questions with a range of scores from 3 to 18, with lower scores indicating a view of personality as changeable.
Hopelessness | Up to 4 weeks after baseline
  Child and parent hopelessness will be assessed via Beck Hopelessness Short Scale, as the primary outcome of Bridging the Gap. This 4-item scale is totaled using the sum of item scores. Scores range from 0-12, with higher scores indicating more hopelessness.

SECONDARY OUTCOMES:
Anxiety Severity | Up to 4 weeks after baseline
  Child anxiety severity will be assessed via SCARED 5-item, as a secondary outcome of Bridging the Gap. This 5-item assessment has scores ranging from 0-10, with higher scores indicating more self-reported anxiety.
Depression Severity | Up to 4 weeks after baseline
  Child and parent depression severity will be assessed via MFQ questionnaire, as a secondary outcome of Bridging the Gap. The MFQ Child version has scores ranging from 0-66, with a higher score indicating more severe depression. The MFQ Parent version has scores ranging from 0-69, with higher score indicating more severe depression.
Psychological distress | Up to 4 weeks after baseline
  Child and parent psychological distress will be assessed via PHQ4 questionnaire, as a secondary outcome of Bridging the Gap. The PHQ4 contains 4 questions, 2 questions relating to depression and 2 questions relating to anxiety, with scores ranging from 0-12. Higher scores on the PHQ4 indicate more severe psychological distress.

CONTACTS AND LOCATIONS:
Overall Officials: Tina Goldstein, PhD, Principal Investigator — University of Pittsburgh; David Brent, MD, Study Director — University of Pittsburgh
Locations (1):
- Children's Community Pediatrics (CCP- Armstrong Kittanning) of Children's Hospital of Pittsburgh of UPMC, Kittanning, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All requests for study data will follow NIMH's data sharing and data use policies. The final completely de-identified dataset(s) will include demographic and clinical data at baseline, and primary and secondary outcomes for all studies, including those funded by the innovation contests. These analytic datasets may also include derived variables with documentation. Our form datasets will include original case report forms, a detailed codebook of variable names, value labels, and programming formats and all study documentation including the protocol and manual of procedures. For descriptive/raw data, study investigators/study staff will upload to NIMH's National Database for Clinical Trials Related to Mental Health Illness (NDCT) on a semi-annual basis all analyzed data being uploaded prior to primary paper publication.
Time Frame: These data will be released to the NDCT soon after each project's "main outcomes" manuscript is accepted for publication
Access Criteria: In addition to public access to the NDCT, data can also be accessed by contacting ETUDES Center investigators.